CLINICAL TRIAL: NCT02033655
Title: A High Protein Weight Loss Intervention for Sarcopenic Obesity in Women
Acronym: POWR-UP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Pork Board (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00050540
Record Dates: First submitted 2014-01-09; First posted 2014-01-13 (Estimated); Last update posted 2019-01-08 (Actual); Status verified 2018-09

CONDITIONS: Weight Loss; Obesity
Keywords: weight loss; older adults; obesity
MeSH Terms: conditions — Weight Loss; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Weight loss high protein (Experimental): Protein supplementation. Subjects follow a calorie-reduction diet for a weight loss of ≥10%, with a high proportion of protein, including substantial amounts of supplemental protein provided as lean beef. Intakes of > 30g of high quality protein will be achieved three times a day by subjects in this group, with all or predominantly all from animal source and 60% of animal protein from pork.
  Interventions: Dietary Supplement: Protein supplementation; Behavioral: Diet counseling and group education lessons
- Weight loss control (Active Comparator): Diet counseling and group education lessons. Subjects follow a calorie-reduction diet for a weight loss of ≥10%.
  Interventions: Behavioral: Diet counseling and group education lessons

INTERVENTIONS:
Dietary Supplement: Protein supplementation — > 30g of high quality protein will be achieved three times a day by subjects in this group, with all or predominantly all from animal source and 60-70% of animal protein from lean pork.
  Arms: Weight loss high protein
Behavioral: Diet counseling and group education lessons — Participants meet once a week for 6 months to participate in group lessons and counseling.

SUMMARY:
The purpose of the trial is to assess the effects of combining regular, generous intakes of high quality protein (primarily from lean pork and other animal source proteins) with calorie restriction on functional status and lean muscle mass in frail, obese, women who participate in a 6 month intervention and 9 month intervention.

DETAILED DESCRIPTION:
Assess the effects of combining regular, generous intakes of high quality protein (primarily from lean pork and other animal source proteins) with calorie restriction on functional status and lean muscle mass in frail, obese, women who participate in a 6 month intervention and 9 month intervention.

For 6 month intervention: Participants will be randomized into one of two study arms: Weight Loss Control (n = 20) subjects follow a calorie-reduced diet for a weight loss or ≥10%; or Weight Loss-High Protein: (n = 40) subjects follow a calorie-reduction diet for a weight loss of ≥10%, with a high proportion of high quality protein at each meal. Intakes of > 30g of high quality protein will be achieved three times a day by subjects in this group, predominantly all from animal sources and 60-70% of animal protein from pork. Subject criteria will include obese (>30 kg/m2) women (≥ 45 yrs.) with mild to moderate functional impairment (by 6 minute walk).

For 9 month intervention: Participants will be randomized into one of two study arms: Weight Loss Control (n = 10) subjects follow a calorie-reduced diet for a weight loss or ≥10%; or Weight Loss-High Protein: (n = 10) subjects follow a calorie-reduction diet for a weight loss of ≥10%, with a high proportion of high quality protein at each meal. Intakes of > 30g of high quality protein will be achieved three times a day by subjects in this group, predominantly all from animal sources and 60-70% of animal protein from pork. Subject criteria will include obese (≥ 30 kg/m2) women (≥ 60 yrs.) with mild to moderate functional impairment (by 6 minute walk).

This is a randomized clinical trial with repeated measurements, with the purpose of assessing change over time for the overall sample and the difference in the High Protein group relative to the Control group with regards to primary outcomes (function and lean body mass). The statistical analyses will proceed chronologically in 3 phases: 1) descriptive analyses that will summarize the distribution of the covariates and dependent variables, 2) bivariate analyses of the association between group membership and the outcome measures, and 3) controlled multivariable analyses, which assess the association between experimental group and the outcomes, controlling for the important covariates.

ELIGIBILITY:
Inclusion Criteria:

* Age 45+ yrs.
* BMI of >30 kg/m2
* Body weight <495 lbs.
* Normal blood chemistries
* Normal renal function
* Primary care physician acknowledgement
* Non-Vegetarian
* Mild to moderate movement impairment

Exclusion Criteria:

* Body weight >495 pounds.
* Current smoker.
* Presence of unstable, acutely symptomatic, or life-limiting illness.
* Positive screen for dementia using Mini-Cog evaluation tool.
* Neurological conditions causing functional or cognitive impairments.
* History of significant weight instability (defined as > 10 pounds weight gain or loss over 6 months prior to study participation).
* Unwillingness or inability to be randomized to any one of two intervention groups, submit to all study testing or continuously participate in a randomly assigned lifestyle intervention program for six months.
* Inability to walk independently.
* Bilateral hip replacements.
* Unable to give consent.
* Unable to complete written recording forms including journals of eating and exercise behaviors.
* Current use of the following medications: monoamine oxidase inhibitors, prescription weight loss medications.
* Primary Care Physician advises against participation.

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2014-03; Primary Completion 2018-08-22 (Actual); Study Completion 2018-08-22 (Actual)

PRIMARY OUTCOMES:
Physical function | Baseline, 4, 6, and 9 months
  Assess the change in 6 minute walk scores at 4, 6, and 9 months
Lean Mass | Baseline, 4, 6, and 9 months
  To assess the change in lean mass at 3 or 4 time points.

SECONDARY OUTCOMES:
Physical Function | Baseline, 4, 6, and 9 months
  To assess the change in SPPB at 4, 6, and 9 months
Weight Loss | Baseline, 4, 6, and 9 months
  To assess the change in body weight at 4, 6, and 9 months
Fat Mass | Baseline, 4, 6, and 9 months
  To assess the change in fat mass at 4, 6, and 9 months

OTHER OUTCOMES:
Change in baseline lipid classes at 6 months | Baseline to 6 months
  Concentrations for lipoprotein classes (VLDL, LDL and HDL particle numbers) were calculated using the LP3 deconvolution algorithm.
Change in baseline lipid subclasses at 6 months | Baseline to 6 months
  Concentrations for lipoprotein (VLDL, LDL, and HDL) subclasses (small, medium and large) were calculated using the LP3 deconvolution algorithm.
Change in baseline lipid participle sizes at 6 months | Baseline to 6 months
  Mean VLDL, LDL and HDL particle sizes were weighted averages derived from the sum of the diameter of each subclass multiplied by its relative mass percentage.
Changes in baseline GlycA at 6 months | Baseline to 6 months
  NMR-measured systemic inflammatory factor and a biomarker of CVD risk.
Change in baseline trimethylamine-N-oxide (TMAO) at 6 months | Baseline to 6 months
  TMAO is a metabolite produced from trimethylamine (TMA) containing nutrients. Nuclear magnetic resonance (NMR) spectroscopy assay was used for quantification of TMAO concentrations.
Change in baseline betaine at 6 months | Baseline to 6 months
  Betaine was measured by 1H-nuclear magnetic resonance (NMR) spectroscopy using a Vantera® NMR Clinical Analyzer (LabCorp, Raleigh, NC).
Change in baseline Lipoprotein Insulin Resistance Index (LP-IR) scores at 6 months | Baseline to 6 months
  LP-IR is a composite metabolomic biomarker that captures the multidimensional effects of insulin resistance on the lipoprotein metabolic chain. It is measured by nuclear magnetic resonance spectroscopy as a weighted score of VLDL, LDL and HDL particle sizes, and their subsets concentrations.
Change in baseline Estimated GFR at 6 months | Baseline to 6 months
  Estimated GFR, which measures renal filtering capacity, is a calculated value based on age, sex, race, and serum creatinine using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation.
Change in baseline fasting glucose at 6 months | Baseline to 6 months
  Level of glucose in the blood after fasting for at least 8 hours

CONTACTS AND LOCATIONS:
Overall Officials: Connie W Bales, PhD, RD, Principal Investigator — Duke University
Locations (1):
- Duke Universtiy Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Derived] Bales CW, Porter Starr KN, Orenduff MC, McDonald SR, Molnar K, Jarman AK, Onyenwoke A, Mulder H, Payne ME, Pieper CF. Influence of Protein Intake, Race, and Age on Responses to a Weight-Reduction Intervention in Obese Women. Curr Dev Nutr. 2017 May 1;1(5):e000703. doi: 10.3945/cdn.117.000703. Epub 2017 Apr 11. PMID 29517074